CLINICAL TRIAL: NCT00057915
Title: A Phase I Study of Active Immunotherapy With CAP-1 (6D) and CMVpp65 Peptide-Pulsed, Autologous Dendritic Cells Produced in the Aastromreplicell Cell Production System in Patients With Stage IV CEA Expressing Malignancies
Brief Title: Vaccine Therapy in Treating Patients With Refractory Stage IV Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Morse, MD, Principal Investigator, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4180; 5910 (Other Grant/Funding Number: NCI); 4180 (Other: Duke IRB)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CEA peptide 1-6D (Experimental): CAP-1(6D) peptide-pulsed, matured, autologous human DC produced by the AastromReplicell™ Cell Production System
  Interventions: Biological: CEA peptide 1-6D

INTERVENTIONS:
Biological: CEA peptide 1-6D — CAP-1(6D) peptide-pulsed, matured, autologous human DC produced by the AastromReplicell™ Cell Production System
  Other Names: carcinoembryonic antigen peptide 1-6D

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells mixed with peptides may make the body build an immune response to kill cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with refractory stage IV cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of administering 1 or 2 courses of vaccination with carcinoembryonic antigen peptide 1-6D (CAP 1-6D)- and CMV pp65 peptide-pulsed autologous dendritic cells in patients with refractory stage IV CEA-expressing malignancies.
* Determine the ability of this regimen to induce CAP 1-6D- and CMV pp65-specific T cells in these patients.
* Determine the antitumor effect of this regimen, in terms of progression-free survival, of these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients undergo leukapheresis and collection of peripheral blood mononuclear cells from which dendritic cells (DC) are generated and pulsed with carcinoembryonic antigen peptide 1-6D (CAP 1-6D) and CMV pp65 peptide. Patients are assigned to 1 of 2 vaccination cohorts.

* Cohort I: Patients receive vaccination with CAP 1-6D-pulsed DC and CMV pp65 peptide-pulsed DC subcutaneously and intradermally every 3 weeks for a total of 4 vaccinations.
* Cohort II: Patients receive vaccinations as in cohort I every 3 weeks for a total of 8 vaccinations.

For both cohorts, a safe dose of the vaccine is defined as the dose at which no more than 1 of 6 patients experiences unacceptable toxicity.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 12 patients (6 per cohort) will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy that is refractory to standard therapy known to have a survival benefit

  * Stage IV disease
* Carcinoembryonic antigen (CEA)-expressing tumor, as evidenced by 1 of the following:

  * Immunohistochemistry with at least 50% of the tumor with at least moderate intensity of staining
  * Peripheral blood CEA greater than 2.5 mg/dL
  * Tumor known to be universally CEA positive (i.e., colon or rectal cancer)
* HLA-A201 positive
* Measurable disease*

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan NOTE: *Histologic or cytologic confirmation is not required for measurable disease restricted to a solitary lesion
* Received at least 1 prior standard chemotherapy regimen known to have a survival benefit
* Previously resected brain metastases allowed provided CT scan or MRI was performed within the past month and shows no metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 6 months

Hematopoietic

* WBC at least 3,000/mm^3
* Hemoglobin at least 9 g/dL (transfusions or red blood cell growth factors [e.g., epoetin alfa] allowed)
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin less than 2.0 mg/dL (unless patient has Gilbert's disease)
* SGOT/SGPT less than 1.5 times upper limit of normal
* No hepatic disease that would preclude study participation
* No viral hepatitis (including chronic hepatitis) by hepatitis B surface antigen and hepatitis C serology

Renal

* Creatinine less than 2.5 mg/dL
* No urinary tract infection

Cardiovascular

* No New York Heart Association class III or IV heart disease

Immunologic

* No history of autoimmune disease, including any of the following:

  * Inflammatory bowel disease
  * Systemic lupus erythematosus
  * Ankylosing spondylitis
  * Scleroderma
  * Multiple sclerosis
* No active acute or chronic infection
* HIV negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious chronic or acute illness that would preclude study participation
* No medical or psychological impediment that would preclude study compliance
* No other malignancy within the past 5 years except nonmelanoma skin cancer, controlled carcinoma in situ of the cervix, or controlled superficial bladder cancer
* No allergy to study vaccine components

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy
* No other concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* At least 6 weeks since prior steroid therapy (except steroids administered as premedication for chemotherapy or contrast-enhanced studies)
* Concurrent hormonal therapy allowed for patients with breast cancer
* No concurrent steroid therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* Recovered from prior therapy
* At least 4 weeks since prior investigational therapy
* At least 4 weeks since other prior therapy
* Any number of prior therapies are allowed
* Concurrent bisphosphonates allowed for bone metastases
* No concurrent immunosuppressive therapy (e.g., azathioprine or cyclosporine)
* No other concurrent experimental therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-09; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  The safety and feasibility of administering one cycle of CAP-1(6D) and CMV pp65 peptide-pulsed, matured, autologous human DC produced by the AastromReplicell™ Cell Production System

SECONDARY OUTCOMES:
Immune response | 12 weeks
  The ability of the epitope pulsed DC to induce CAP-1(6D) and CMV pp65-specific T cells

CONTACTS AND LOCATIONS:
Overall Officials: Herbert K. Lyerly, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States